CLINICAL TRIAL: NCT06496945
Title: Assessing the Impact of DAy Programs on Individuals Living with Dementia and Their Family/friend Caregivers (AIDA-DemCare)
Brief Title: Assessing the Impact of DAy Programs on Individuals Living with Dementia and Their Family/friend Caregivers
Status: Recruiting | Type: Observational
Sponsor: York University (Other)
Collaborators: Carswell Family Foundation (Unknown); Alzheimer Society of York Region (Unknown)
Responsible Party: Principal Investigator, Matthias Hoben, Associate Professor, Helen Carswell Chair in Dementia Care, York University
Other Study IDs: 563198
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Adult Day Programs; Continuing Care; Old Age; Dementia; Family/Friend Caregivers
Keywords: Adult day programs; Older adults; Program evaluation; Cohort studies; Health administrative data
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Day program attendees & caregivers: Older adults (65+ years), living with a diagnosis of dementia in the community, and attending an adult day program in the Calgary Health Zone (Alberta), Interior Health Region (British Columbia), Winnipeg Regional Health Authority (Manitoba), or York Region (Ontario). Each older adult's primary caregiver (i.e., the person most involved with and informed about the care of the older adult) will also be recruited.
  Interventions: Other: Adult day program use
- Non-attendees & caregivers: Older adults (65+ years), living with a diagnosis of dementia in the community in the Calgary Health Zone (Alberta), Interior Health Region (British Columbia), Winnipeg Regional Health Authority (Manitoba), or York Region (Ontario), with an initial Resident Assessment Instrument - Home Care (RAI-HC) completed, but who are not attending a day program. Each older adult's primary caregiver (i.e., the person most involved with and informed about the care of the older adult) will also be recruited.
  Interventions: Other: Other community care (non-attendees)

INTERVENTIONS:
Other: Adult day program use — Day program use patterns will be determined, using Latent Class Analysis. Three continuous variables will be categorized as low, low-moderate, high-moderate, high, using sample distribution quartiles: (1) Time between first RAI-HC assessment and first attendance of a day program, (2) average number of hours of day program attendance (i.e., total number of hours spent in a day program divided by the number of times attended), and (3) total number of days a person attended a day program.
  Groups: Day program attendees & caregivers
Other: Other community care (non-attendees) — Any publicly funded continuing care services in the community, other than adult day programming (e.g., home care, in-home respite). Community care participants will be propensity score matched with day program participants, using RAI-HC variables on day program eligibility (to ensure similarity of non-attendees to day program attendees). Matching variables will include: physical functioning, cognition, behavioural symptoms, bladder/bowel continence, availability of a caregiver, and caregiver distress. The investigators will also include variables on health and social characteristics (e.g., age, sex, type/duration of publicly funded community care received before the matching index date, deprivation indices).
  Groups: Non-attendees & caregivers

SUMMARY:
This study seeks to understand the effects of adult day programs on older adults, especially those with dementia, and their caregivers. A prospective cohort study will be conducted in the Canadian provinces of Alberta, British Columbia, Manitoba, and Ontario. Participants will be (1) older adults with dementia who attend a day program, and their caregivers, and (2) older adults with dementia in the community who do not attend a day program, and their caregivers. The objectives are to (1) evaluate the effects of day programs on attendee and caregiver outcomes, and (2) compare day program use patterns, attendee and caregiver social identities, day program characteristics, and day program outcomes between the 4 provinces, and (3) to explore what attendee and caregiver social identities and day program characteristics are associated with study outcomes, and with day program attendance/non-attendance.

DETAILED DESCRIPTION:
Adult day programs provide critical supports to both, older adults with dementia in the community, and their family/friend caregivers. This is critical because ensuring high-quality care in the community for as long as possible, and avoiding or delaying facility-based continuing care are key priorities of individuals with dementia, their caregivers, and healthcare systems. While 61% of the 597,000 Canadians with dementia live in the community, about 10% of newly admitted nursing home residents have relatively low care needs that could be met in the community with the right supports. Caregivers to individuals with dementia (most of whom are women) provide more care hours per week (26 vs 17) than caregivers to older adults without dementia, are more likely to experience distress (45% vs 26%), and a caregiver's risk of distress is 1.6 times higher if the individual in need of care exhibits behavioural problems. However, research on the effectiveness of day programs is inconsistent. Generally, the methodological quality of studies is poor, and we especially lack Canadian research and research on individuals with multiple, intersecting vulnerabilities. Our research objectives are:

1. To evaluate the association of day program exposure with primary outcomes (better quality of life of attendees and caregivers), and secondary outcomes (better mental health of attendees and caregivers, increased time to admission to congregate care, slower cognitive and physical decline of attendees, lower rates of attendees' and caregivers' emergency room registrations, hospital admissions, and days in hospital)
2. To compare day program use patterns, attendee and caregiver social identities, day program characteristics, and day program outcomes between the 4 provinces
3. To explore what attendee and caregiver social identities, and day program characteristics are associated with primary and secondary outcomes, and with day program attendance/non-attendance

In this prospective, cross-provincial cohort study (York Region, Ontario; Interior Health, British Columbia; Calgary, Alberta; Winnipeg, Manitoba), a total of 1,000 day program attendees with dementia (250 per region), plus their primary caregivers will be recruited. A comparison group of 2,000 non-attendees with dementia and their caregivers will be created. Participants' longitudinal health administrative data will be combined with repeated (baseline and after 1 and 2 years) surveys to include critical variables not routinely collected by healthcare systems (e.g., quality of life, social identities). Primary study outcomes are quality of life of the person with dementia and their caregiver. Secondary study outcomes include mental health of individuals with dementia and caregivers, cognitive and physical decline of individuals with dementia, time to admission to congregate care, and system-level rates of emergency room registrations, hospital admissions, and days in hospital (including alternative level of care) of individuals with dementia and caregivers. Using a day program survey, we will also assess day program characteristics (e.g., number of spaces, staffing, programming). Using general estimating equations and time-to-event models, these outcomes will be compared between groups of day program exposure (no, low, medium, high). Models will be adjusted for community-based services (e.g., home care, respite care), day program characteristics, social identities of older adults and caregivers, time since day program admission, and other older adult and caregiver characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (65+ years) with a diagnosis of dementia, who live in the community, and either attend an adult day program (cohort 1), or receive continuing care in the community with an initial RAI-HC assessment completed (cohort 2)
* Primary caregiver (i.e., most involved with and informed about the care) of an eligible older adult

Exclusion Criteria:

* Older adults with or without dementia who do not receive any community-based continuing care service
* Day program attendees or community care recipients who do not have a diagnosis of dementia or who are younger than 65 years
* Secondary caregivers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study focuses on community care systems in the Calgary Health Zone (Alberta), Interior Health Region (British Columbia), Winnipeg Regional Health Authority (Manitoba), and York Region (Ontario). All of these regions assess day program eligibility using comparable processes, criteria, and assessments (i.e. RAI-HC). There are 89 publicly subsidized day programs in Alberta (~3,300 spaces), 95 (~1,500 spaces) in British Columbia, 70 (~1,000 spaces) in Manitoba, and 300 (~6,000 spaces) in Ontario. The numbers of individuals with dementia in the community are ~32,000 in Alberta, ~47,000 in British Columbia, ~11,000 in Manitoba, ~153,000 in Ontario.
  The yearly average number of completed RAI-HC assessments is ~20,000-30,000 in Alberta, ~34,000-39,000 in British Columbia, and ~10,000 in Manitoba. The estimated number of day program attendees is >20,000/year (>200,000 within the study period), each with multiple assessments.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Older adult quality of life (self-report) | Baseline (Jan-Mar 2025), and after 1 and 2 years
  For older adults who can self-report (cognitive performance scale score of < 3), the DEMQOL will be completed as part of an older adult survey (administered as a standardized interview). The DEMQOL is a tool to assess dementia-specific quality of life, but according to the tool developers, there is no spelled-out version of this acronym. Each of 28 items is rated on a scale from 1 to 4 and items are summed for an overall score from 28 to 112 (higher scores = better quality of life).
Older adult quality of life (proxy-report) | Baseline (Jan-Mar 2025), and after 1 and 2 years
  For all older adults (including those who can or cannot self-report), the DEMQOL-Proxy will be completed as part of a caregiver survey (administered as a standardized interview). The DEMQOL is a tool to assess dementia-specific quality of life, but according to the tool developers, there is no spelled-out version of this acronym. Each of 31 items is rated on a scale from 1 to 4 and summed for an overall score from 31 to 124 (higher scores = better quality of life).
Caregiver quality of life | Baseline (Jan-Mar 2025), and after 1 and 2 years
  As part of our caregiver survey, the C-DEMQOL will be completed (administered as a standardized interview). The C-DEMQOL is a tool to assess quality of life of caregivers to persons with dementia, but according to the tool developers, there is no-spelled out version of this acronym. Each of 30 items is rated on a scale from 1 to 5 and summed for an overall score from 30 to 150 (higher scores = better quality of life).

SECONDARY OUTCOMES:
Older adult mental health | Baseline (Jan-Mar 2025), and after 1 and 2 years
  The Neuro Psychiatric Inventory (NPI) will be completed as part of a caregiver survey (administered as a standardized interview). The NPI measures the severity (0 = not present, 1 = mild, 2 = moderate, 3 = severe) of each of 12 neurological and behavioural symptoms of dementia. Symptoms include delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances, and appetite and eating abnormalities. Scores are summed for an overall score between 0 and 36 (with higher scores indicating more and more severe symptoms).
Caregiver distress | Baseline (Jan-Mar 2025), and after 1 and 2 years
  The Neuro Psychiatric Inventory (NPI) will be completed as part of a caregiver survey (administered as a standardized interview). In addition to the severity of the 12 neurological and behavioural symptoms of dementia mentioned above, the NPI also measures the level of distress each of these symptoms causes to the caregiver (from 0 = not distressing at all to 5 = extreme or very severe). Scores are summed for an overall score between 0 and 60 (with higher scores indicating more severe distress).
Caregiver symptoms of depression | Baseline (Jan-Mar 2025), and after 1 and 2 years
  The 10-item Center for Epidemiologic Studies Depression Scale, Short Form (CES-D10) will be completed as part of a caregiver survey (administered as a standardized interview). A cut-point of ≥ 10 will be used to identify clinically significant depressive symptoms
Caregiver symptoms of anxiety | Baseline (Jan-Mar 2025), and after 1 and 2 years
  The 7-item Generalized Anxiety Disorder scale (GAD-7) will be completed as part of a caregiver survey (administered as a standardized interview). A cut-point of ≥ 8 will be used to identify clinically significant symptoms of anxiety.
Presence or absence of physical decline among older adults | Baseline (Jan-Mar 2025), and after 1 and 2 years
  Change in physical functioning will be captured, using the validated RAI-HC Activities of Daily Living Hierarchy (ADLh) scale. The scale ranges from 0 (no impairment) to 6 (maximum impairment), and the outcome will be dichotomous, indicating any increase (versus no change or a decrease) between the previous and follow up measurement in this scale. RAI-HC data are routinely collected by the healthcare system, and we will request data for each participant at each of the specified measurement time points.
Presence or absence of cognitive decline among older adults | Baseline (Jan-Mar 2025), and after 1 and 2 years
  Change in cognition will be captured, using the validated RAI-HC Cognitive Performance Scale (CPS). The scale ranges from 0 (no impairment) to 6 (maximum impairment), and the outcome will be dichotomous, indicating any increase (versus no change or a decrease) between the previous and follow up measurement in this scale. RAI-HC data are routinely collected by the healthcare system, and we will request data for each participant at each of the specified measurement time points.
Older adult time to admission to a continuing care home | From date of home care admission until the date of admission to a continuing care home or loss to follow up (i.e., death, move out of province), whichever came first, assessed up to 2.5 years (between baseline and 2-year follow up)
  Data will come from provincial continuing care registries, which document the start date of any publicly funded continuing care service a person receives, the end date of this service, and the type of service. The outcome will be the time between a person's first RAI-HC assessment and admission to a continuing care home (i.e., an assisted living home or nursing home).
Older adult emergency room registrations | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  The National Ambulatory Care Report System (NACRS) captures all emergency department visits and diagnoses. The outcome will be the yearly average number of a person's emergency department visits.
Caregiver emergency room registrations | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  The National Ambulatory Care Report System (NACRS) captures all emergency department visits and diagnoses. The outcome will be the yearly average number of a person's emergency department visits.
Older adult hospital stays | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  The Discharge Abstract Database (DAD) includes information on all inpatient hospital stays, including diagnoses and length of stay. The outcome will be the yearly average number of a person's hospital stays.
Caregiver hospital stays | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  The Discharge Abstract Database (DAD) includes information on all inpatient hospital stays, including diagnoses and length of stay. The outcome will be the yearly average number of a person's hospital stays.
Older adult primary care provider visits | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  Care provider claims data includes health service claims submitted for payment by primary care providers (e.g., general practitioners, nurse practitioners, geriatricians, geriatric psychiatrists, neurologists, therapists). The outcome will be the yearly average number of a person's primary care provider visits.
Caregiver primary care provider visits | 1 and 2 years after the baseline data collection (which is estimated to be carried out Jan-Mar 2025)
  Care provider claims data includes health service claims submitted for payment by primary care providers (e.g., general practitioners, nurse practitioners, geriatricians, geriatric psychiatrists, neurologists, therapists). The outcome will be the yearly average number of a person's primary care provider visits.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hoben, Dr rer medic, Principal Investigator — York University
Locations (4):
- Canada (4):
  - Edmonton and Calgary Health Zones, Edmonton & Calgary, Alberta
  - Interior Health Region, Multiple, British Columbia
  - Winnipeg Regional Health Authority, Winnipeg, Manitoba
  - York Region, Multiple, Ontario

IPD SHARING:
Plan to Share IPD: No
The data collected in this study include identifiable, sensitive healthcare variables. Therefore, we are required by provincial regulations and by our ethics boards to keep and analyze the data in a secure, encrypted, and firewall protected virtual data environment. Only persons who meet regional and provincial confidentiality requirements will be allowed to access the data. Data access can be requested with the principal investigator of this study and eligibility will be determined on an individual basis.

REFERENCES:
- [Derived] Hoben M, Ubell A, Maxwell CJ, Allana S, Doupe MB, Symonds-Brown H, Hogan DB, Daly T, Tate KC, Wagg A, Nguyen H, Berta W, Bethell J, Caspar S, Goodarzi Z, McGrail K, Cummings GG, Rowe M, Kay K, Kostyk P, Lazaruk K, MacLean B, Mann J, Prescott K. Assessing the impact of day programs on individuals living with dementia and their family/friend caregivers (AIDA-DemCare): protocol of a prospective cohort study combined with a qualitative evaluation. BMC Public Health. 2025 Aug 19;25(1):2846. doi: 10.1186/s12889-025-23896-6. PMID 40830776